CLINICAL TRIAL: NCT06285747
Title: A Correlational Study: Breast Cancer-Related Chest Wall Lymphedema, Quality of Life, and Shoulder Function
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-004117; NCI-2024-01191 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-004117 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients complete questionnaires and undergo chest wall and breast lymphedema measurements by clinical assessment and using the Delfin Moisture Meter D Compact and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study evaluates how swelling in the chest following breast cancer treatment may affect patients' quality of life and shoulder function.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if there is a correlation to Delfin Moisture Meter Compact D reading and quality of life as measured by the LymQOL-midline.

II. Determine if there is a correlation to Delfin Moisture Meter Compact D reading and DASH measure of shoulder function.

III. Determine how the presence of chest wall lymphedema as determined by physical exam may affect an individual's quality of life as measured by the LymQOL-midline assessment.

IV. Determine how the presence of chest wall lymphedema as determined by physical exam may shoulder function on the effected side, as measured by the Disabilities of the Arm, Shoulder, and Hand questionnaire.

OUTLINE: This is an observational study.

Patients complete questionnaires and undergo chest wall and breast lymphedema measurements by clinical assessment and using the Delfin Moisture Meter D Compact and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Women of any age with diagnosis of any type of breast cancer

  * Breast cancer on unilateral or bilateral side
  * Surgical intervention for treatment of breast cancer

Exclusion Criteria:

* Previous shoulder injury or known shoulder limitation on affected side

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who have undergone surgical intervention for treatment of breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Chest wall lymphedema | Baseline
  Assessed using the the MoistureMeterD Compact, handheld device by Delfin Technologies.
Quality of life - Limb Lymphoedema Quality of Life (LymQOL) | Baseline
  Assessed using the Limb Lymphoedema Quality of Life (LymQOL) Tool, a patient reported outcome measure comprised of 20 questions. Responses for questions 1-19 are: not at all, a little, quite a bit, a lot, or N/A with free-text fields for participants to include examples. Question 20 is answered on a 1-10 scale. Higher scores generally indicate better quality of life.
Disability of the shoulder - Disabilities of the Arm, Shoulder and Hand (DASH) | Baseline
  Assessed using the Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire. Questions are answered with a scale of 1-5 with varying values assigned to the numbers (e.g., not at all, slightly, moderately, quite a bit, extremely). Higher scores indicate greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Kayla A. Van Der Weerd, PT, DPT, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials